CLINICAL TRIAL: NCT00223574
Title: Long-Term Effect of Altering the Source or Amount of Dietary Carbohydrate in Type 2 Diabetes
Brief Title: Canadian Trial of Dietary Carbohydrates in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 44205
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: Control - high carbohydrate, high glycemic index foods
Drug: high carbohydrate, low glycemic index foods
Drug: low carbohydrate, high monounsaturate fat foods

SUMMARY:
A long-term low carbohydrate, high monounsaturated fat diet, compared to a high carbohydrate, low glycemic index diet, results in more rapid progression of diabetes; i.e. increased fasting glucose and glycated hemoglobin, reduced beta-cell function and insulin sensitivity and increased free fatty acids. The deleterious effects of a high carbohydrate diet on plasma lipids are only temporary and do not persist beyond 6 months. A long-term high carbohydrate, low glycemic index diet, compared to a high carbohydrate, high glycemic index diet, improves glycemic control and beta-cell function

ELIGIBILITY:
Inclusion Criteria:

* male or non-pregnant/non-lactating females with type 2 diabetes treated by diet alone
* age 53-75y
* body mass index 25-40kg/m^2 (Caucasian) or 23-40kg/m^2 (other)
* HbA1c <=130% of upper limit of normal of local hospital lab

Exclusion Criteria:

* use of any hypoglycemic or anti-hyperglycemic drug within 6 months of randomization
* major cardiovascular event or major surgery within 6 months of randomization
* serum triglycerides >10mmol/L
* presence of other major debilitating disorder such as liver disease, renal failure or cancer
* presence of gastrointestinal disorder or use of drug which is likely to alter gastrointestinal motility or nutrient absorption
* use of oral steroids
* substance or alcohol abuse
* simultaneous participation in another clinical trial
* allergy or intolerance to more than one of wheat, barley, corn, oats, potato, legumes, nuts, psyllium, olives, avocado or canola
* unwilling or unable to follow the protocol and/or give informed consent
* subjects planning to be on holiday for more than 8 weeks in a row or a total of 12 weeks in the year in locations to which they will not take study food

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168
Dates: Start 2002-01; Study Completion 2004-10

PRIMARY OUTCOMES:
glycated hemoglobin

SECONDARY OUTCOMES:
Body weight
waist circumference
occurrence of diet failure
fasting glucose
fasting C-reactive protein
fasting lipids (total, HDL and LDL cholesterol and triglcyerides)
fasting apolipoproteins A1 and B100
fasting free fatty acids
fasting short chain fatty acids
plasma glucose and insulin 30, 60 and 120min after 75g oral glucose
insulin sensitivity (HOMA)
beta-cell function (30min-fasting insulin)/(30min-fasting glucose)
metabolic profile (glucose, insulin, triglycerides and FFA during 8h profile)
quality of life
gastrointestinal symptoms
diet satisfactio

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, MD, PhD, Principal Investigator — University of Toronto/St. Michael's Hospital
Locations (5):
- Canada (5):
  - Clinical Trials Centre, Edmonton, Alberta
  - St. Joseph's Health Centre, London, Ontario
  - St. Michael's Hosptial, Toronto, Ontario
  - Hotel Dieu, Montreal, Quebec
  - Centre Universitaire de Sante de l'estrie, Sherbrooke, Quebec